CLINICAL TRIAL: NCT00646230
Title: A Phase I Study of Intravenous (Emulsion) Fenretinide in Children With Recurrent or Resistant Neuroblastoma
Brief Title: N2004-03: Intravenous Fenretinide in Treating Young Patients With Recurrent or Resistant Neuroblastoma
Acronym: IV Fenretinide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nant Operations Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Nant Operations Center, NANT Operations Center, Children's Hospital Los Angeles
Organization: Children's Hospital Los Angeles (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000584267; P01CA081403 (NIH); N2004-03 (Other: NANT Consortium)
Record Dates: First submitted 2008-03-27; First posted 2008-03-28 (Estimated); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Fenretinide; Chromatography, High Pressure Liquid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm of CIV infusion of emulsion 4-HPR (Experimental): Single arm study of continuous intravenous infusion (CIV) of emulsion 4-HPR
  Interventions: Drug: fenretinide; Other: high performance liquid chromatography; Other: pharmacological study

INTERVENTIONS:
Drug: fenretinide
Other: high performance liquid chromatography
Other: pharmacological study

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fenretinide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I trial is studying the side effects and best dose of intravenous fenretinide in treating young patients with recurrent or resistant neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of fenretinide when given as a continuous intravenous infusion in young patients with recurrent and/or resistant neuroblastoma.
* To define the toxicities of this drug in these patients.
* To determine the plasma pharmacokinetics of this drug in these patients.

Secondary

* To determine the response rate in patients treated with this drug.
* To determine the bioavailability of fenretinide in normal peripheral blood mononuclear cells as a surrogate marker for drug bioavailability to tumor tissue.

OUTLINE: This is a multicenter study.

Patients receive fenretinide IV continuously over 120 hours on days 0-4. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for pharmacokinetic analysis by high performance liquid chromatography.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of neuroblastoma either by histological confirmation and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines

  * Differentiating ganglioneuroblastoma allowed

    * No histological evidence only of ganglioneuroma by tumor biopsy or bone marrow biopsy
* High-risk disease meeting at least one of the following criteria:

  * Recurrent/progressive disease at any time
  * Refractory disease (i.e., less than a partial response to front-line therapy that included ≥ 4 courses of chemotherapy)
  * Persistent disease after at least a partial response to front-line therapy (i.e., still has residual disease by MIBG, CT/MRI, or bone marrow biopsy)

    * Biopsy of at least one residual site demonstrating viable neuroblastoma required (tumor by bone marrow morphology is considered adequate documentation of disease)
* Measurable disease meeting at least one of the following criteria:

  * Measurable tumor on MRI or CT scan, defined as at least one unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan

    * For patients with persistent disease, a biopsy* of bone marrow or bone or soft tissue site must have demonstrated viable neuroblastoma
  * MIBG scan with positive uptake at a minimum of one site

    * For patients with persistent disease, a biopsy* of a MIBG positive site must have demonstrated viable neuroblastoma
  * Bone marrow with tumor cells seen on routine morphology (not by NSE staining only) of bilateral aspirate and/or biopsy of one bone marrow sample NOTE: *If the lesion was irradiated, the biopsy must have been done at least 4 weeks after completion of radiotherapy
* No CNS parenchymal or meningeal-based lesions

  * Skull-based tumor lesions with or without intracranial extension are allowed provided there are no neurologic signs or symptoms or hydrocephalus related to the lesion
  * Patients with a history of complete surgical resection of CNS lesions are eligible provided there is no evidence of CNS lesions by MRI or CT scan at study entry
  * Patients with a history of CNS lesions must be off corticosteroid therapy for CNS lesions for ≥ 4 weeks

PATIENT CHARACTERISTICS:

* Performance status 0-2
* Life expectancy ≥ 2 months
* ANC ≥ 500/mm³
* Platelet count ≥ 50,000/mm³ (transfusion independent)
* Hemoglobin ≥ 8.0 g/dL (transfusion independent)
* Serum creatinine ≤ 1.5 times normal for age
* Total bilirubin ≤ 1.5 times normal for age
* ALT and AST ≤ 3 times normal for age
* Serum triglycerides < 300 mg/dL
* Serum calcium < 11.6 mg/dL
* Lipase normal for age
* PT/PTT ≤ 1.5 times upper limit of normal for age (without fresh frozen plasma support; vitamin K allowed)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to, during, and for 2 months after completion of study treatment
* LVEF ≥ 55% by ECHO or MUGA scan OR fractional shortening ≥ 27% by ECHO
* No EKG abnormality
* No dyspnea at rest or requirement for oxygen
* No hematuria and/or proteinuria > 1+ on urinalysis
* No known history of allergy to egg products
* No known history of allergy to soy bean oil
* No skin toxicity > grade 1 per CTCAE v3
* Seizure disorder allowed if seizures are controlled on anticonvulsants and the anticonvulsant(s) is not contraindicated
* Known genetic, metabolic, or psychiatric conditions, or other ongoing serious medical issues must be approved by the study chair prior to study registration

PRIOR CONCURRENT THERAPY:

* Recovered from all prior chemotherapy, immunotherapy, or radiotherapy
* More than 3 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosoureas) and/or biologic therapy without stem cell support
* More than 7 days since prior hematopoietic growth factors
* No prior radiotherapy to the only site of measurable disease unless there has been subsequent disease progression at that site or a biopsy of that site showed viable neuroblastoma ≥ 4 weeks after completion of radiotherapy
* Prior CNS irradiation allowed
* At least 2 weeks since prior small field (focal) radiotherapy
* At least 6 weeks since prior large field radiotherapy (i.e., total-body irradiation, craniospinal radiotherapy, whole abdominal or total lung radiotherapy, or radiotherapy to > 50% of marrow space)
* At least 56 days since prior myeloablative autologous stem cell transplantation
* At least 4 weeks since prior myelosuppressive therapy with stem cell support
* At least 6 weeks since prior MIBG therapy
* Prior oral fenretinide therapy allowed
* At least 3 weeks since prior retinoid therapies
* No prior organ transplantation
* No prior myeloablative allogeneic stem cell transplantation unless stem cells were from an identical twin sibling
* No concurrent systemic corticosteroids, including corticosteroids for emesis control

  * Concurrent inhaled corticosteroids for asthma control or steroids for metabolic deficiency states allowed
* Concurrent palliative radiotherapy allowed provided the irradiated sites will not be used to measure response
* No concurrent parenteral intralipids
* No other concurrent chemotherapy or immunomodulating agents
* No concurrent drugs suspected of causing pseudotumor cerebri, including tetracycline, nalidixic acid, nitrofurantoin, phenytoin, sulfonamides, lithium, or amiodarone
* No concurrent vitamin A, C, or E supplements (except as part of routine total parenteral nutrition [TPN] supplements or as part of a single daily standard dose of oral multivitamin supplement)
* No concurrent medications that may potentially act as modulators of intracellular ceramide levels or ceramide cytotoxicity, sphingolipid transport, or p-glycoprotein (MDR1) or MDR1 drug/lipid transporters, including cyclosporine or analogue, verapamil, tamoxifen or analogue, ketoconazole, chlorpromazine, mifepristone (RU486), indomethacin, or sulfinpyrazone
* No other concurrent anticancer agents
* No concurrent herbal supplements or other alternative therapy medications
* No concurrent anti-arrhythmia or inotropic cardiac medications

Ages: 0 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2006-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To define the toxicities of intravenous emulsion 4-HPR given on this schedule. | Adverse events, clinically significant changes in lab results or vitals will be captured throughout the duration of the study.
  Adverse events, clinically significant changes in lab results or vitals will be captured throughout the duration of the study.
To determine the maximum tolerated dose of intravenous emulsion 4-HPR given as a continuous intravenous infusion (CIV) for five days (120 hours) every three weeks in children with recurrent and/or resistant neuroblastoma. | Tolerability of drug will be assessed throughout the study.
To determine the plasma pharmacokinetics of intravenous emulsion 4-HPR given on this schedule. | Pharmacokinetic Profile of Fenretinide - blood levels to be measured in Cycle #1 D0 Hr0, Hrs 6, 12, 24, 36, 48, 72, 96, 120 and end of infusion, then +2 hrs, +48 hrs post infusion. Cycle #2 D1 Hr0 (pre-infusion), then +48 hrs, at the end of infusion.

SECONDARY OUTCOMES:
To determine the response rate to intravenous emulsion 4-HPR in patients with recurrent and/or resistant neuroblastoma within the confines of a Phase I study. | Disease response will be assessed at baseline, End of Cycle #2, End of Cycle #6 and every 4 weeks thereafter.
  Response will be measured utilizing any of the following;CT scan, MRI, MIBG scan, Bone Marrow, Urine Catecholamines
To determine the bioavailability to tumor cells of 4-HPR delivered as an intravenous emulsion in normal peripheral blood mononuclear cells (PBMC) as a tumor cell surrogate tissue. | Assessed Cycle #1 D0 Hr0, D2, +48hrs after start of infusion and C#2 one time for patients >20kg.
To describe the results of the five gene Five-gene TaqMan® Low Density Array (TLDA) assay for neuroblastoma tumor cells in the bone marrow done at timepoints when bone marrow response is being evaluated by morphology during this therapy. | Assessed at the end of Cycle #2 & Cycle #6 and then every 4 cycles therafter.

CONTACTS AND LOCATIONS:
Overall Officials: Barry J. Maurer, MD, PhD, Study Chair — Texas Tech University Health Sciences Center
Locations (13):
- United States (12):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - University of Chicago Comer Children's Hospital, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Morgan Stanley Children's Hospital of New York-Presbyterian, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Texas Children's Cancer Center and Hematology Service at Texas Children's Hospital, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada